CLINICAL TRIAL: NCT03459573
Title: Fit-One: A Randomized Waitlist Controlled Trial Evaluating the Effect of One Drop and Fitbit on Diabetes and Pre-diabetes Outcomes
Brief Title: Fit-One: A Trial Evaluating the Effect of One Drop and Fitbit on Diabetes and Pre-diabetes Outcomes
Acronym: Fit-One
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Chandra Osborn, PhD, MPH (Industry)
Responsible Party: Sponsor-Investigator, Chandra Osborn, PhD, MPH, VP, Health & Behavioral Informatics, Informed Data Systems, Inc.
Organization: Informed Data Systems, Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Fit-One
Record Dates: First submitted 2018-02-20; First posted 2018-03-09 (Actual); Last update posted 2019-08-09 (Actual); Status verified 2019-08

CONDITIONS: Diabetes Mellitus, Type 2; Diabetes Mellitus, Type 1; PreDiabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus, Type 1; Prediabetic State

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (7):
- T2D: One Drop with Fitbit Ionic (Active Comparator)
  Interventions: Behavioral: One Drop | Experts On Track
- T2D: One Drop without Fitbit Ionic (Active Comparator)
  Interventions: Behavioral: One Drop | Experts On Track
- T2D: Waitlist Control (No Intervention)
- T1D: One Drop with Fitbit Ionic (Active Comparator)
  Interventions: Behavioral: One Drop | Experts On Call
- T1D: One Drop without Fitbit Ionic (Active Comparator)
  Interventions: Behavioral: One Drop | Experts On Call
- PD: One Drop with Fitbit Charge 2 (Active Comparator)
  Interventions: Behavioral: One Drop | Experts Revive
- PD: One Drop without Fitbit Charge 2 (Active Comparator)
  Interventions: Behavioral: One Drop | Experts Revive

INTERVENTIONS:
Behavioral: One Drop | Experts On Track — Participants with T2D will use One Drop's digital therapeutics solution (app, meter, and 'On Track' in-app coaching) for 3 months
  Arms: T2D: One Drop with Fitbit Ionic; T2D: One Drop without Fitbit Ionic
Behavioral: One Drop | Experts On Call — Participants with T1D will use One Drop's digital therapeutics solution (app, meter, and 'On Track' in-app coaching) for 3 months
  Arms: T1D: One Drop with Fitbit Ionic; T1D: One Drop without Fitbit Ionic
Behavioral: One Drop | Experts Revive — Participants with pre-diabetes will use One Drop's digital therapeutics solution (app, meter, and 'Revive' in-app coaching) for 3 months
  Arms: PD: One Drop with Fitbit Charge 2; PD: One Drop without Fitbit Charge 2

SUMMARY:
The Fit-One trial involves three prospective, randomized waitlist-controlled studies. These studies evaluate the effects of One Drop's digital therapeutics solution with and without Fitbit devices on the social cognitive, behavioral, and health outcomes of people with diabetes. Fit-One is being tested on adults with type 1 diabetes (T1D) of all weights, and adults with type 2 diabetes (T2D) or pre-diabetes that are overweight or obese (BMI ≥ 25).

DETAILED DESCRIPTION:
Sub-study 1 (T2D). Eligible participants (N=300) with T2D, an A1c above 7.0% and Body Mass Index (BMI) ≥ 25 will be randomized to one of three groups. Participants assigned to group 1 (n=100) get One Drop's digital therapeutics solution (app, meter, and 'On Track' in-app coaching) and a Fitbit Ionic smartwatch and are asked to use both for 3 months. Participants assigned to group 2 (n=100) get One Drop's digital therapeutics solution and are asked to use it for 3 months. After 3 months, group 2 gets a Fitbit Ionic smartwatch. Finally, participants assigned to group 3 (n=100) are asked to manage their diabetes without an app, coach, or activity tracker for 3 months. After 3 months, group 3 gets One Drop's digital therapeutics solution (app, meter, and 'On Track' in-app coaching) and a Fitbit Ionic smartwatch (n=100).

Sub-study 2 (T1D). Eligible participants (N=100) with T1D and an A1c above 7.0% will be randomized to one of two groups. Participants assigned to group 1 (n=50) get One Drop's digital therapeutics solution (app, meter, and 'On Call' in-app coaching) and a Fitbit Ionic smartwatch and are asked to use both for 3 months. Participants assigned to group 2 (n=50) get One Drop's digital therapeutics solution and are asked to use it for 3 months. After 3 months, group 2 gets a Fitbit Ionic smartwatch.

Sub-study 3 (Pre-diabetes). Eligible participants (N=100) with pre-diabetes, an A1c between 5.7-6.4% and a BMI ≥ 25 will be randomized to one of two groups. Participants assigned to group 1 (n=50) get One Drop's digital therapeutics solution ('Revive' in-app coaching) and a Fitbit Charge 2 and are asked to use both for 3 months. Participants assigned to group 2 (n=50) get One Drop's digital therapeutics solution and are asked to use it for 3 months. After 3 months, group 2 gets a Fitbit Charge 2.

ELIGIBILITY:
Inclusion Criteria:

* 18-75 years of age
* U.S. residency and mailing address
* Self-reported diagnosis of T1D, T2D, or pre-diabetes
* For people with a diabetes diagnosis, diagnosed for 1+ years
* For people with a diabetes diagnoses, self-reported A1c ≥ 7.0% (later confirmed with a mail-in A1c laboratory test)
* For people with a pre-diabetes diagnoses, self-reported A1c 5.7-6.4% (later confirmed with a mail-in A1c laboratory test)
* For people with T2D or pre-diabetes, BMI ≥ 25
* Owns and uses an iPhone or Android phone
* No cardiovascular problems
* No neuromuscular problems
* No orthopedic problems
* Doctor is ok with increased physical activity
* English-speaking
* Naïve to One Drop's digital therapeutics solution
* Naïve to all Fitbit products

Exclusion Criteria:

* Currently pregnant or planning to become pregnant during the trial period
* Cannot read or write in English
* Currently in a diabetes education or coaching program
* Previously downloaded the One Drop | Mobile app
* Owns or previously used Fitbit products

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2018-02-23 (Actual); Primary Completion 2018-08-31 (Actual); Study Completion 2019-12-01 (Estimated)

PRIMARY OUTCOMES:
Hemoglobin A1c | 3 months
  Within- and between-group changes in central lab-assessed A1c measured at baseline and 3 months.

SECONDARY OUTCOMES:
Weight | 3 months (12 months for Sub-study 3)
  Within- and between-group changes in self-reported weight measured at baseline and follow-up(s). In sub-study 3, the Fitbit Aria Wi-Fi scale will assess weight at baseline, 4, 8, and 12 months post-baseline.
Healthcare Utilization | 3 months (12 months for Sub-study 3)
  Within- and between-group change in the number of emergency room visits and hospitalizations. This will be assessed with two self-reported items that ask: (1) How many times have you gone to the emergency room in the past 3 months? and (2) How many times have you been admitted to the hospital in the past 3 months?
Diet | 3 months (12 months for Sub-study 3)
  Within- and between-group diet changes. The Summary of Diabetes Self-Care Activities (SDSCA) general and specific diet subscales will measure self-reported 7-day diet behavior at baseline and follow-up(s). The One Drop app will collect daily and weekly diet behavior that's manually entered during the trial period.
Physical Activity | 3 months (12 months for Sub-study 3)
  Within- and between-group activity changes. The SDSCA exercise subscale will measure self-reported 7-day exercise behavior at baseline and follow-up(s). The One Drop app will also collect daily and weekly activity that's manually-entered and/or passively-collected via HealthKit, Google Fit, or a Fitbit tracker or smartwatch during the trial period.
Medication Adherence | 3 months (12 months for Sub-study 3)
  Within- and between-group medication adherence changes. The SDSCA medications subscale will measure self-reported 7-day medication adherence at baseline and follow-up(s). The One Drop app will also collect daily and weekly medication taking that's manually-entered into the app during the trial period.
Self-Monitoring of Blood Glucose | 3 months
  Within- and between-group self-monitoring of blood glucose (SMBG) changes. The SDSCA SMBG subscale will measure self-reported 7-day SMBG at baseline and follow-up. During the trial period, the One Drop app will collect daily and weekly SMBG that's manually-entered and/or passively-collected via the One Drop | Chrome Bluetooth-connected glucose meter.

OTHER OUTCOMES:
Health-related Productivity | 3 months (12 months for Sub-study 3)
  Within- and between-group change in health-related productivity. The Work Productivity and Activity Impairment measure will measure self-reported work productivity (absenteeism, presenteeism and daily activities) at baseline and follow-up(s).
Health-related Quality of Life | 3 months (12 months for Sub-study 3)
  Within- and between-group change in health-related quality. The CDC HRQOL-14 will measure self-reported health-related quality of life at baseline and follow-up(s).
Life Satisfaction | 3 months (12 months for Sub-study 3)
  Within- and between-group change in life satisfaction. Cantril's Self-Anchoring Ladder of Life Satisfaction will measure self-reported life satisfaction at baseline and follow-up(s).

CONTACTS AND LOCATIONS:
Locations (1):
- One Drop, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Herman WH, Rothberg AE. Prevalence of Diabetes in the United States: A Glimmer of Hope? JAMA. 2015 Sep 8;314(10):1005-7. doi: 10.1001/jama.2015.10030. No abstract available. PMID 26348749
- [Background] Tuomilehto J, Lindstrom J, Eriksson JG, Valle TT, Hamalainen H, Ilanne-Parikka P, Keinanen-Kiukaanniemi S, Laakso M, Louheranta A, Rastas M, Salminen V, Uusitupa M; Finnish Diabetes Prevention Study Group. Prevention of type 2 diabetes mellitus by changes in lifestyle among subjects with impaired glucose tolerance. N Engl J Med. 2001 May 3;344(18):1343-50. doi: 10.1056/NEJM200105033441801. PMID 11333990
- [Background] Diabetes Prevention Program (DPP) Research Group. The Diabetes Prevention Program (DPP): description of lifestyle intervention. Diabetes Care. 2002 Dec;25(12):2165-71. doi: 10.2337/diacare.25.12.2165. PMID 12453955
- [Background] Marathe PH, Gao HX, Close KL. American Diabetes Association Standards of Medical Care in Diabetes 2017. J Diabetes. 2017 Apr;9(4):320-324. doi: 10.1111/1753-0407.12524. No abstract available. PMID 28070960
- [Background] Krass I, Schieback P, Dhippayom T. Adherence to diabetes medication: a systematic review. Diabet Med. 2015 Jun;32(6):725-37. doi: 10.1111/dme.12651. Epub 2015 Jan 9. PMID 25440507
- [Background] Green AJ, Bazata DD, Fox KM, Grandy S; SHIELD Study Group. Health-related behaviours of people with diabetes and those with cardiometabolic risk factors: results from SHIELD. Int J Clin Pract. 2007 Nov;61(11):1791-7. doi: 10.1111/j.1742-1241.2007.01588.x. Epub 2007 Sep 20. PMID 17887992
- [Background] Peyrot M, Rubin RR, Lauritzen T, Snoek FJ, Matthews DR, Skovlund SE. Psychosocial problems and barriers to improved diabetes management: results of the Cross-National Diabetes Attitudes, Wishes and Needs (DAWN) Study. Diabet Med. 2005 Oct;22(10):1379-85. doi: 10.1111/j.1464-5491.2005.01644.x. PMID 16176200
- [Background] Cadmus-Bertram LA, Marcus BH, Patterson RE, Parker BA, Morey BL. Randomized Trial of a Fitbit-Based Physical Activity Intervention for Women. Am J Prev Med. 2015 Sep;49(3):414-8. doi: 10.1016/j.amepre.2015.01.020. Epub 2015 Jun 10. PMID 26071863
- [Background] Vangeepuram N, Williams N, Constable J, Waldman L, Lopez-Belin P, Phelps-Waldropt L, Horowitz CR. TEEN HEED: Design of a clinical-community youth diabetes prevention intervention. Contemp Clin Trials. 2017 Jun;57:23-28. doi: 10.1016/j.cct.2017.03.010. Epub 2017 Mar 23. No abstract available. PMID 28344183
- [Background] Baye E, Menon K, de Courten MP, Earnest A, Cameron J, de Courten B. Does supplementation with carnosine improve cardiometabolic health and cognitive function in patients with pre-diabetes and type 2 diabetes? study protocol for a randomised, double-blind, placebo-controlled trial. BMJ Open. 2017 Sep 1;7(9):e017691. doi: 10.1136/bmjopen-2017-017691. PMID 28864708
- [Background] Coughlin SS, Hatzigeorgiou C, Anglin J, Xie D, Besenyi GM, De Leo G, Stewart J, Wilkins T. Healthy lifestyle intervention for adult clinic patients with type 2 diabetes mellitus. Diabetes Manag (Lond). 2017;7(2):197-204. PMID 28794802
- [Background] Gow ML, Baur LA, Johnson NA, Cowell CT, Garnett SP. Reversal of type 2 diabetes in youth who adhere to a very-low-energy diet: a pilot study. Diabetologia. 2017 Mar;60(3):406-415. doi: 10.1007/s00125-016-4163-5. Epub 2016 Nov 26. PMID 27889809
- [Background] Diaz KM, Krupka DJ, Chang MJ, Peacock J, Ma Y, Goldsmith J, Schwartz JE, Davidson KW. Fitbit(R): An accurate and reliable device for wireless physical activity tracking. Int J Cardiol. 2015 Apr 15;185:138-40. doi: 10.1016/j.ijcard.2015.03.038. Epub 2015 Mar 4. No abstract available. PMID 25795203
- [Derived] Osborn CY, Hirsch A, Sears LE, Heyman M, Raymond J, Huddleston B, Dachis J. One Drop App With an Activity Tracker for Adults With Type 1 Diabetes: Randomized Controlled Trial. JMIR Mhealth Uhealth. 2020 Sep 17;8(9):e16745. doi: 10.2196/16745. PMID 32540842